CLINICAL TRIAL: NCT02273999
Title: Pulsed Electromagnetic Fields for Postoperative Pain: a Randomized Controlled Clinical Trial in Patients Undergoing Mandibular Third Molar Extraction
Brief Title: Pulsed Electromagnetic Fields for Postoperative Pain: a Linical Trial in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova, School of Dental Medicine (Other)
Responsible Party: Principal Investigator, Stefano Sivolella, Clinical Faculty department of oral surgery, University of Padova, School of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2976P
Record Dates: First submitted 2014-10-15; First posted 2014-10-24 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Pain; Oral Surgery; Third Molar Extraction
Keywords: pulsed electromagnetic fields; post operative morbidity; third molar; extraction; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (no device) (No Intervention): No devices were delivered after third molar tooth extraction
- Placebo group (Inactivated device) (Placebo Comparator): Inactivated devices were delivered after third molar tooth extraction
  Interventions: Device: RecoveryRx™
- Test (activated device) (Experimental): Activated devices were delivered after third molar tooth extraction
  Interventions: Device: RecoveryRx™

INTERVENTIONS:
Device: RecoveryRx™ — Appliance of the device after surgery
  Other Names: Pulsed electromagnetic fields
  Arms: Placebo group (Inactivated device); Test (activated device)

SUMMARY:
This randomized clinical trial was designed to assess the clinical efficacy of Pulsed electromagnetic field PEMF delivered with a wearable device in terms of postoperative pain and quality of healing after mandibular third molar extraction.

The sample included 120 patients undergoing unilateral mandibular third molar extraction. The devices were positioned over the area corresponding to the extraction site and wearers were asked to keep them in place for 7 days. All patients were asked to record pain (on a visual analog scale [VAS]), hours of wearing the device (groups T and P), and any use of analgesics. At 7 days, healing complications (dehiscence, tumefaction, pus, local lymphadenopathy, pain on palpation, postoperative bleeding, alveolitis) were recorded blindly.

DETAILED DESCRIPTION:
Introduction: Pulsed electromagnetic field (PEMF) therapy is a noninvasive method for delivering pulsed radiofrequency energy to tissues to treat postoperative pain and edema. This randomized clinical trial was designed to assess the clinical efficacy of PEMF delivered with a wearable device in terms of postoperative pain and quality of healing after mandibular third molar extraction.

Materials and methods: The sample included 120 patients undergoing unilateral mandibular third molar extraction. At the end of the surgical procedure, patients were randomly assigned to a test (T) or placebo (P) group and fitted with enabled or disabled PEMF devices, respectively, or to a control (C) group not fitted with a PEMF device. The devices were positioned over the area corresponding to the extraction site and wearers were asked to keep them in place for 7 days. All patients were asked to record pain (on a visual analog scale [VAS]), hours of wearing the device (groups T and P), and any use of analgesics. At 7 days, healing complications (dehiscence, tumefaction, pus, local lymphadenopathy, pain on palpation, postoperative bleeding, alveolitis) were recorded blindly.

ELIGIBILITY:
Inclusion Criteria:

* patients who needs third molar extraction,
* good oral hygiene,
* no contraindications to treatment.

Exclusion Criteria:

* age under 14 years;
* poor oral hygiene (plaque index less then 20%);
* contraindications for surgery (or anesthesia);
* infectious or systemic diseases;
* immunosuppressant therapy;
* pregnancy or breastfeeding;
* mental disorders.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Visual Analog scale | up to day 7 post intervention

SECONDARY OUTCOMES:
Quality of healing | day 7 post intervention
  The quality of healing will be measured by scoring the presence of the following: dehiscence, tumefaction, pus, local lymphadenopathy, pain on palpation, postoperative bleeding, alveoli tis will be recorded blindly for each patients. Frequency of complications (per patients) at 7 days. Numerical values and p-values of comparisons will be recorded.